CLINICAL TRIAL: NCT01435629
Title: Open-label, Multicenter, Observational, Non-intervention Study to Retrospectively Evaluate the Efficacy of Norditropin® (Adult Height) in Patients With Achondroplasia/Hypochondroplasia Enrolled in the GH-1941 Study [Follow-up Survey]
Brief Title: A Survey Collecting Data on Adult Height in Patients With Achondroplasia Treated With Somatropin
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: GH-3907; U1111-1121-7729 (Other: WHO); JapicCTI-111622 (Other: JAPIC)
Record Dates: First submitted 2011-09-14; First posted 2011-09-16 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Genetic Disorder; Achondroplasia
MeSH Terms: conditions — Genetic Diseases, Inborn; Achondroplasia | interventions — Human Growth Hormone

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Norditropin®
  Interventions: Drug: somatropin

INTERVENTIONS:
Drug: somatropin — Dosage and administration to be prescribed by the physician as a result of a normal clinical practice.

SUMMARY:
This study is conducted in Japan. The aim of the study is to evaluate the efficacy of somatropin (Norditropin®) on adult height (cm) in patients with achondroplasia / hypochondroplasia enrolled in the GH-1941 study (NCT01516229).

ELIGIBILITY:
Inclusion Criteria:

* Patients who were enrolled in the GH-1941 study (1997 to 2006) and expected to theoretically reach the adult height within the study period

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients enrolled in the GH-1941 study (NCT01516229) expected to achieve the adult height by 2015 and available for follow-up by the investigator
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2012-11-22 (Actual); Primary Completion 2015-12-04 (Actual); Study Completion 2015-12-04 (Actual)

PRIMARY OUTCOMES:
To collect change data of adult height (cm) of patients treated with Norditropin® and evaluate the long-term efficacy | At year 1, 2, 3, 4, and 5 after the patient has reached adult height or is 18 of age

SECONDARY OUTCOMES:
To monitor the patients to see if they undergo lower limb lengthening | At year 1, 2, 3, 4, and 5 after the patient has reached adult height or is 18 of age

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Tokyo, Japan

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com